CLINICAL TRIAL: NCT03317054
Title: Prevalence of Pathologic Gambling in the Workforce: a Cross-sectional Study in Brittany, France
Acronym: PJPAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PJPAP
Record Dates: First submitted 2017-08-07; First posted 2017-10-23 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Behavior and Behavior Mechanisms
Keywords: Gambing; occupational health services; psychosocial risks
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Introduction: To date, very few studies about links between work and addictive disorders concern behavioral addictive disorders such as gambling. Such behaviours may be adaptative strategy for unsatisfied workers. The common physiopathology of addictive disorders allows us to hypothesize that it is possible that such troubles at work could promote gambling. Our aim was to evaluate the prevalence of gambling among workers and its links with work.

Patients and methods: We performed a descriptive cross-sectional monocentric study among all workers who consulted one physician between November 2016 and April 2017, from an occupational health service in Brittany, France. The first step was to ask whether they have gambled during the last year and if it was related to their occupation. The second step was a screening for risky gamblers (using the "Lie or Bet" questionnaire) among these and then to assess more precisely the severity (using the Indice Canadien du Jeu Excessif, ICJE questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* all employees coming in consultation in occupational medicine, between the 2016-11-01 and the 2017-04-30, with the investigator, having given their consent and replied to the questionnaires were included.

Exclusion Criteria:

* Employees who did not speak the French language and those who refused to participate in the study were excluded. The number of refusals to participate and their reason were identified by the investigator. In addition, for employees who came to consult several times during the collection period, we only included the data from the first visit, in order to avoid overrepresentation.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: employees coming in consultation in occupational medicine, between the 2016-11-01 and the 2017-04-30
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Gambling prevalence | 6 month

SECONDARY OUTCOMES:
link between workand gambling | 6 month
type of game | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Santé au travail en cornouaille, Quimperlé, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No